CLINICAL TRIAL: NCT06376422
Title: Sterile Allogeneic Spongioflex® Allograft as Partial Meniscal Replacement After Incomplete Meniscal Loss, an Investigator-initiated Low Interventional Trial.
Brief Title: Sterile Allogeneic Spongioflex® Allograft as Partial Meniscal Replacement After Incomplete Meniscal Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sven Behrendt (Other)
Responsible Party: Sponsor-Investigator, Sven Behrendt, principal investigator, Privatpraxis für Knie- und Schulterchirurgie
Organization: Privatpraxis für Knie- und Schulterchirurgie (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU-CT-2023-508271-36-00
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Meniscus Lesion
Keywords: meniscus deficiency; partial meniscus replacement; Spongioflex®; Allograft; International Knee Documentation Committee (IKDC) Score; Knee Injury and Osteoarthritis Outcome Score (KOOS); Visuelle Analogskala (VAS) Score; Extrusion; magnetic resonance imaging (MRI)
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Masking Description: no masking, patient decides which group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spongioflex® (Experimental): As for any surgical procedure, the patient receives an antibiotic shot non-interventional medicinal product (NIMP) just before surgery. The patient will be arthroscopically treated via the arthroscopic portal with implantation of a demineralized bone block (IMP: Spongioflex ®, appropriate size (DIZG gGmbH, Berlin, Germany)) as a partial meniscus substitute. The block will be adapted to the defect size and secured with 2-4 inside-out sutures (Etibond 0, Ethicon, Somerville, NJ). No dosing, the IMP has no systemic effect. The surgery (Intervention) will last between 60-90 minutes. The hospital stay is between 2-3 days after surgery. Follow-up visits: at the end of the hospital stay, after 6 weeks, after 6, 12 and 24 months and after 5 years for the operated group.
  Interventions: Procedure: Spongioflex®
- non-operated (Other): no surgical treatment, no antibiotic shot, no visit at the end of the hospital stay, and no visit after 6 weeks. Follow-up visits after 6, 12 and 24 months and after 5 years.
  Interventions: Other: non-operated

INTERVENTIONS:
Procedure: Spongioflex® — partial meniscal replacment during surgery, follow-up visits at the end of hospital stay and after 6 weeks, MRI evaluation and questionnaires after 6, 12, 24 and 60 months.
  Arms: Spongioflex®
Other: non-operated — no surgery, MRI evaluation and questionnaires follow-up after 6, 12, 24 and 60 months
  Arms: non-operated

SUMMARY:
The goal of this clinical trial is to learn if partial meniscal replacement can prevent or postpone total meniscal replacement, in adult patients (female/male) with partial meniscal loss. The main questions it aims to answer are:

* Can partial meniscal replacement improve knee function?
* Can partial meniscal replacement prevent/postpone total meniscal replacement/knee prothesis? Researchers will compare the results of the operated group with patients not willing to be operated but with partial meniscal loss to see if the operation improves knee function.

Participants will be operated and have to attend follow-up visits with MRI after 6 months up to 5 years after surgery.

DETAILED DESCRIPTION:
The menisci consist of fibrocartilage. They are partially (laterally more than medially) mobile parts of the joint surfaces and compensate for the incongruence of the femur and tibia. They reduce the joint pressure on the tibial plateau and the femoral condyles and help to stabilize the joint. Due to this biomechanical relevance, the partial loss of the meniscus leads to arthritic changes in long term. Suturing the torn meniscus is increasingly becoming the focus of knee surgery. Degenerative torn menisci have a significantly poorer prognosis with regard to healing than traumatically torn menisci (e.g. meniscus damage associated with a cruciate ligament tear).

Indications for partial meniscus replacement are symptomatic, degenerative, and irreparable damage to the medial and lateral meniscus, possibly with early osteoarthritis of the compartments, as well as partial loss of the meniscus in the event of anterior knee instability in young, active patients, in which case simultaneous reconstruction of the anterior cruciate ligament should be performed. A prerequisite for a good clinical result after partial meniscus replacement is a stable knee without malalignment in the coronal plane. Partial meniscus replacement is not suitable in the case of axial deviation and knee instability, patients older than 60 years, advanced chondromalacia and degenerative changes in the affected compartment, an extension deficit of more than 3° compared to the opposite side or a knee flexion of less than 125°. Inflammatory arthritis or synovial inflammation of the knee and a Body Mass Index (BMI) greater than 30 kg/m² are additional exclusion criteria.

Williams et al. 2007 could show, that 5 years after partial removal of the medial or lateral meniscus, despite an excellent functional result, 64% of patients showed medial and 33% lateral cartilage damage on magnetic resonance imaging (MRI). This study highlights the considerable delay with which the symptoms occur despite already detectable arthritic changes.

Englund et al. were able to show in a study that patients developed osteoarthritis significantly more frequently over a period of 30 months if they had meniscus damage than if they did not. Englund et al. detected tibiofemoral osteoarthritis in 27% of patients 15 years after partial meniscus removal compared to 10% in a control group that had not undergone surgery.

In the case of incomplete meniscus loss, where the peripheral rim is sufficiently intact, defect filling is the only way to restore the lost substance and function of the meniscus. In the past, an implant made of bovine collagen (Collagen Meniscus Implant (CMI), Stryker) or an artificial meniscus made of polyurethane (Actifit, 2med) was often used. The CMI has been withdrawn from the market by the manufacturer, so that no biological treatment alternative exists.

Schenk et al. were able to show in a recent study for the CMI, consisting of bovine collagen that, despite a significant improvement in pain and function, the CMI is subject to a progressive shrinkage process over time. The studies mentioned above make it clear that partial replacement of the meniscus is necessary if preservation by meniscus suturing is no longer possible to prevent or postpone arthritic changes.

In the investigator-initiated study on which this application is based, a novel implant made from demineralized allogenic human cancellous bone (Spongioflex®, DIZG gGmbH Berlin) is to be implanted into the meniscus defect of the recipient knee. This transplant has sponge-like properties and therefore facilitates the ingrowth of cells from the surrounding meniscus. The investigational medicinal product (IMP, Spongioflex®) is de-calcified and demineralized, it is hard, when dry, but soft when wet. In the knee the conditions are wet, thus it stays soft. It is pliable (Fig1) and can be easily sutured.

Figure 1: Spongioflex®

The manufacturer (Deutsches Institut für Zell-und Gewebeersatz (DIZG gGmbH)) did a study of cell ingrowth on Spongioflex®. They describe that ingrowth of cells on Spongioflex® was observed after 28 days and these cells do not ossify.

Scotti et al. summarizes 2013 the knowledge in respect to meniscal repair as follows:

"In the last decade, striving for optimal restoration of meniscal tissue, the orthopedic surgeon's armamentarium has been enriched by the use of biocompatible meniscus scaffold and meniscal allograft transplantation". "However, despite promising short-term results, none of the current strategies have demonstrated regeneration of a functional, long-lasting meniscal tissue and re-establishment of a proper knee homeostasis in the meniscectomised knee". "The rationale for using a cell-free biomaterial to replace part of the meniscus is based on repopulation of the scaffold by the host cells recruited from the synovium and the meniscal remnants, and subsequent tissue ingrowth which renders this approach cell-based after implantation. A mandatory prerequisite is the absence of both knee instability and malalignment".

This section of the paper of Scotti et al. describes exactly the need for a restoration of the meniscus. Furthermore it defines exactly the features of a scaffold:

"A biomaterial used as scaffold for meniscus tissue engineering purposes should present many features. In particular, the ideal meniscal scaffold should be (i) "cell-instructive", promoting cell differentiation and proliferation if cell-seeded, or cell migration if cell-free; (ii) "biomimetic", mimicking architecture, tribology and mechanical features of the native meniscus; (iii) resilient and resistant to withstand mechanical forces acting in the joint while cells produce extra cellular matrix (ECM); (iv) biocompatible, not evoking any foreign-body reaction also with its degradation products; (v) slowly biodegradable allowing to be gradually replaced by biologic tissue; (vi) open, with high porosity, allowing diffusion of nutrients and catabolic substances; and (vii) easy to handle, to be sutured and to be implanted by the surgeon".

Pereira et al. describes that a meniscal implant, either for partial or total replacement should:

"provide the biomechanical properties but also the biological features to replace the loss of native tissue. Moreover, these approaches include possibilities for patient-specific implants of correct size and shape".

Spongioflex® fulfils all these demands described by Dabaghi et al., Scotti et al. and Peirera et al. and it can be adapted in size and shape and thus is in the moment the optimal choice for partial meniscal replacement.

Dickerson et al. describes that "the scaffold must have a high fluid conductance, concomitant with high porosity…. Porosity allows more rapid cell incorporation along the surface and through the thickness of the scaffold, promoting integration with the host tissue.". "The scaffold must guide cells to regenerate all four zones of the tissue structure".

This is the case of Spongioflex® it is porose and can guide cells. Scotti et al. proposes 2013 to use CMI for partial meniscal regeneration, but this product is retracted from the market by now and they describe already the shrinking of the transplant. Knee stability and an aligned knee are a requisite for the study proposed. Dickerson et al. shows that new fibrocartilage tissue is formed on the demineralized end of the allograft. Results of Credille et al. support these findings. It will not be ossified again. Smith et al. describes that "demineralized cancellous bone sponges are Food and Drug Administration-approved and commercially available products that have the potential to provide biologic and biomechanical augments for rotator cuff healing. The sponge can act as a scaffold for cellular attachment and proliferation" .

Credille et al. showed in a recent publication that a biphasic interpositional cancellous allograft (BioEnthesis; Sparta BioPharma, Inc., Madison, NJ) can be used for rotator cuff repair. The allograft is "a porous scaffold for endogenous biological factor migration and thus potentially address the lack of enthesis recapitulation at the rotator cuff repair interface… while the demineralized layer supports soft-tissue ingrowth while acting as a "sponge" to hold bone marrow elements at the repair site".

The group around Prof. Moroder from the Charité has used Spongioflex® for glenoid repair. They describe that the transplant does not calcify again. The glenoid is also no bony structure. They used the same product in non-bone structures and could show successful restoration of the glenoid.

Sundar et al. describes that the use demineralized bone matrix increased fibrocartilage when used for augmentation of rotator cuff repair. The used graft (Spongioflex®) provides a scaffold for cell migration of meniscal cells from neighbouring parts of the meniscus. The intended study will show that this kind of allograft is suitable for partial meniscal replacement because it allows cell migration and has enough porosity to allow fluid conductance. [24] As described by Wildemann et al. sufficient growth factors are remaining in the demineralized bone matrix (Spongioflex®) to support new fibrocartilage formation. Scotti et al. underlines the importance of growth factors for meniscal regeneration.

In summary from the literature, it can be concluded, that Spongioflex® is an attractive scaffold for partial meniscal repair because it is fully biological, it still has fibrocartilage inductive factors, allows cell migration, fluid conductivity, resists biomechanical forces, does not provoke immunoreactivity, it is adaptable in size and can easily be sutured. Partial meniscus replacement is an established surgical treatment for patients who have undergone partial meniscus removal, to lead to the ingrowth of cells and the regeneration of meniscus-like tissue.

The purpose of this investigator-initiated trial is to evaluate whether the novel graft can prevent/reduce the disadvantages of the previously used replacement materials and shows better results than the group of patients, which were not operated. Since there is currently no alternative made of biological material to this product, this investigator-initiated trial is of great medical and economic importance. The otherwise following arthrosis or knee prosthesis implantation (TKA) could be prevented or at least postponed. Initial clinical results are promising.

An important and sensitive parameter for assessing the postoperative function of the meniscus is the MRI image. Genovese et al. 2007 were able to show in a categorization/classification which magnetic resonance image can be expected in the case of successful incorporation. Several studies have shown that the known clinical knee scores (Lysholm, nternational Knee Documentation Committee (IKDC), Knee Injury and Osteoarthritis Outcome Score (KOOS), Visual Analogue Scale (VAS) pain) improve significantly after successful ingrowth of the meniscus implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male and female) with:
2. Partial loss of portions of the

   * lateral meniscus and lateral joint line pain OR
   * medial meniscus and medial joint line pain
3. sufficient standing of the peripheral rim, so that the procedure can be performed
4. Age: 18-60 years
5. signed written informed consent to the study and to provide the scientific data in pseudonymized form

Exclusion Criteria:

1. The presence of anterior cruciate ligament insufficiency which is not resolved by reconstruction of the anterior cruciate ligament within 16 weeks after partial meniscal implantation.
2. Axial deviation (>2° varus or valgus)
3. realignment osteotomy not performed within 12 weeks
4. advanced cartilage damage (grade III according to ICRS) and osteoarthrosis in the affected compartment (grade III according to Kellgren and Lawrence [33])
5. Extension deficit of more than 3° compared to the opposite side or a knee flexion of less than 125°
6. inflammatory arthritis or synovitis on the treated knee
7. BMI greater than 30 kg/m²
8. <18 years, >60 years
9. Chronic pain patients
10. only for patients who will be operated:

    1. with increased anaesthesiologic risk, e.g., with known or predicted difficult airway
    2. with increased risk of bleeding
    3. with increased risk of infection
    4. with necrotic, infected, or poorly perfused host sides
    5. history of allergic reactions
    6. acute hypersensitivity reactions to the IMP or any of its excipients
    7. pregnant woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of the procedure | 5 years
  Improvement of knee function after surgery compared to the non-operated group and compared to pre-surgery scores.
Improvement of International Knee Documentation Committee (IKDC) score (between 0 and 100, the higher the better) | 5 years
  Improvement of IKDC Score after surgery compared to the non-operated group and compared to pre-surgery scores.
Improvement of Knee Injury and Osteoarthritis Outcome Score (KOOS) score (between 0 and 100, the higher the better) | 5 years
  Improvement of KOOS score after surgery compared to the non-operated group and compared to pre-surgery scores.
Improvement of Visual Analogue Scale (VAS) Pain Score (between 0 and 10, the lower the better) | 5 years
  Improvement of VAS Pain score after surgery compared to the non-operated group and compared to pre-surgery scores.

SECONDARY OUTCOMES:
Safety of the patient (adverse events (AE) and serious adverse events (SAE)) | 5 years
  Type, frequency and severity of treatment-related AEs and SAEs
Efficacy of the procedure, progression to osteoarthrosis | 5 years
  How many patients show a progression of osteoarthrosis up to total knee arthroplasty (TKA)?
Menuiscus size | 5 years
  size of meniscus ((mm), depends on location, gender and height of patient), after 6 weeks, 6 and 12 months (for operated patients) and after 2 and 5 years, comparison between the operated and the non-operated group
extrusion of meniscus | 5 years
  extrusion of meniscus (yes/no, no extrusion is better) after 6 weeks, 6 and 12 months (for operated patients) and after 2 and 5 years, comparison between the operated and the non-operated group
Size of meniscal extrusion | 5 years
  Size of meniscal extrusion ((mm) the smaller the better) after 6 weeks, 6 and 12 months (for operated patients) and after 2 and 5 years, comparison between the operated and the non-operated group
Patient satisfaction | 5 years
  The scale of patient satifaction is: very pleased, pleased, not pleased, very unsatisfied in the operated group after 2 and 5 years, which will be asked in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sven Behrendt, MD, Principal Investigator — Privatpraxis für Knie- und Schulterchirurgie
Locations (1):
- Privatpraxis für Knie und Schulterchirurgie, Dortmund, Germany

IPD SHARING:
Plan to Share IPD: No
no sharing plan

REFERENCES:
- [Background] Behrendt S. MRI follow up of bilateral partial meniscal substitution with a demineralized bone block. A case report. Radiol Case Rep. 2022 Oct 27;18(1):21-26. doi: 10.1016/j.radcr.2022.09.091. eCollection 2023 Jan. PMID 36324835

DOCUMENTS (1):
  • Study Protocol (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT06376422/Prot_000.pdf